CLINICAL TRIAL: NCT02308085
Title: A Study Evaluating the Pregnancy Outcomes and Safety of Interrupting Endocrine Therapy for Young Women With Endocrine Responsive Breast Cancer Who Desire Pregnancy
Brief Title: Pregnancy Outcome and Safety of Interrupting Therapy for Women With Endocrine Responsive Breast Cancer
Acronym: POSITIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Alliance for Clinical Trials in Oncology (Other); Canadian Cancer Trials Group (Network); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 48-14 / BIG 8-13; Alliance A221405 (Other: Alliance for Clinical Trials in Oncology); NCIC CTG MAC.18 (Other: NCIC Clinical Trials Group)
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Early Breast Cancer
Keywords: Premenopausal; endocrine responsive; Breast; Pregnancy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endocrine therapy interruption (Experimental): Endocrine therapy interruption after having completed between ≥ 18 months and ≤ 30 months.
  Interventions: Other: Endocrine therapy interruption

INTERVENTIONS:
Other: Endocrine therapy interruption — 3 months wash-out between treatment interruption and pregnancy attempt. Up to 2 years interruption to allow pregnancy, delivery, breastfeeding or failure to conceive.
  Endocrine therapy resumption. Completion of full duration of endocrine therapy according to individual risk, institutional policy or patient's preference.

SUMMARY:
The best available evidence suggests that pregnancy after breast cancer does not increase a woman's risk of developing a recurrence from her breast cancer. In particular, the most recent data suggest that this is the case also in women with a hormone receptor-positive breast cancer. There is also no indication of increased risk for delivery complications or for the newborn. The aim of the study is to investigate if temporary interruption of endocrine therapy, with the goal to permit pregnancy, is associated with a higher risk of breast cancer recurrence.The study aims also to evaluate different specific indicators related to fertility, pregnancy and breast cancer biology in young women. A psycho-oncological companion study on fertility concerns, psychological well-being and decisional conflicts will be conducted in interested Centers.

DETAILED DESCRIPTION:
Recent decades have witnessed a delay in childbearing for a variety of reasons including cultural, educational, and professional. As a consequence, breast cancer in young women often occurs before the completion of reproductive plans. Infertility has a significant impact on quality of life, resulting in substantial distress in younger women with breast cancer and influencing treatment decisions in a consistent proportion of patients.The best available evidence suggests that pregnancy after breast cancer does not increase a woman's risk of developing a recurrence.For women desiring pregnancy after a breast cancer, 5-10 years of endocrine therapy may substantially reduce the chance of conception; however, a shorter duration of endocrine therapy in this population has not been studied in a prospective manner.

Birth outcome after breast cancer has not been shown to be different from that of the normal population, but increased risks of delivery complications, cesarean section, preterm birth and low birth weight have been reported.

Endocrine agents are potentially teratogenic: taking into account their median half-life, waiting 3 months after their interruption before attempting conception is considered safe.

The limited evidence available on breastfeeding after breast cancer reports successful lactation from the treated breast in approximately 30% of women without detrimental effect on survival. No prospective definitive data are available.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 42 years at enrollment.
* Has received adjuvant endocrine therapy (SERM alone, GnRH analogue plus SERM or AI) for ≥18 months but ≤30 months for early breast cancer.

Note: Patients who have received neo/adjuvant endocrine treatment within a clinical trial and patients who have received pharmaco-prevention are eligible.

* The adjuvant endocrine therapy must have stopped within 1 month prior to enrollment.
* Patient wishes to become pregnant. Note: Patients who have undergone oocyte/embryo/ovarian tissue cryopreservation at breast cancer diagnosis and/or have a previous history of assisted reproductive technology (ART) are eligible.
* Breast cancer for which patient is receiving endocrine therapy must have been histologically-proven stage I-III, endocrine-responsive (i.e., estrogen and/or progesterone receptor positive, according to local definition of positive, determined using immunohistochemistry (IHC)), and treated with curative intent.

Note:

* Patients with synchronous bilateral invasive breast cancer (diagnosed histologically within 2 months) are eligible.
* Patient with invasive breast cancer or synchronous bilateral invasive breast cancer (diagnosed histologically within 2 months) during pregnancy are eligible.
* Patients with BRCA1/2 mutations are eligible.
* Patients could have received neo/adjuvant chemotherapy, or other systemic therapy (e.g., neo/adjuvant HER2-targeted therapy) according to institutional policy and patient's desire.
* Patient must be premenopausal at breast cancer diagnosis, as determined locally and documented in patient record.
* Patient must be without clinical evidence of loco-regional and distant disease, as evaluated according to institutional assessment standards and documented in the patient record.
* Written informed consent (IC) for trial participation must be signed and dated by the patient and the investigator prior to enrollment.
* Written consent to biological material submission, indicating the patient has been informed of and agrees to tissue and blood material use, transfer and handling, must be signed and dated by the patient and the investigator prior to any procedures specific for this trial.
* The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.
* Patient must be accessible for follow-up.

Exclusion Criteria:

* Post-menopausal patients at BC diagnosis, as determined locally.
* History of hysterectomy, bilateral oophorectomy or ovarian irradiation.
* Patients with current local, loco-regional relapse and/or distant metastatic breast cancer.
* Patients with a history of prior (ipsi- and/or contralateral) invasive BC.
* Patients with previous or concomitant non-breast invasive malignancy.
* Exceptions are limited exclusively to patients with the following previous malignancies, if adequately treated: basal or squamous cell carcinoma of the skin, in situ non-breast carcinoma, contra- or ipsilateral in situ breast carcinoma, stage Ia carcinoma of the cervix.
* Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical disorder that would interfere with the patient's safety.
* Patients with a history of noncompliance to medical treatments and/or considered potentially unreliable.
* Patients with psychiatric, addictive, or any disorder that would prevent compliance with protocol requirements.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 518 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer free interval (BCFI) | From enrollment until the first invasive BC event, assessed up to 14 years
  Kaplan-Meier Analysis

SECONDARY OUTCOMES:
Information on Menstruation recovery and pattern | Up to 24 months after enrollment
  Menstrual diary
Pregnancy rate (determined by pregnancy test) | Up to 24 months after enrollment
  Pregnancy test
Pregnancy outcome | Up to 33 months after enrollment
  Labor and delivery Information, full term pregnancy, caesarean section, abortion, miscarriage, ectopic, stillbirth rates.
Offspring outcome | Up to 33 months after enrollment
  Collect information on preterm birth, low birth weight, births defects rates.
Breastfeeding pattern | Up to 36 months after enrollment
  Analysis of pattern e.g Duration, use of ipsilateral breast if previous breast conservation, side exclusivity
Use of assisted reproductive Technology (ART) | Up to 24 months after enrollment
  ART use will be tabulated
Distant recurrence-free interval (DRFI) | Time from enrollment in the study to the first breast cancer recurrence in a distant site, assessed up to 14 years
  Kaplan-Meier Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Pagani, MD, Study Chair — Oncology Institue of Southern Switzerland (IOSI)
Locations (211):
- United States (103):
  - Cedars Sinai Medical Centre, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Sharp Memorial Hospital, San Diego, California
  - University of Colorado Cancer Centre - Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University - Yale Cancer Centre, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newport, Delaware
  - Regional Hematology Oncology Practice Associates, Newport, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - OnCare Hawaii Inc - POB I, Honolulu, Hawaii
  - Queen's Medical Centre, Honolulu, Hawaii
  - OnCare Hawaii-Kuakini, Honolulu, Hawaii
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group - Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - NorthShore University Health System - Glenbrook Hospital, Glenview, Illinois
  - NorthShore Unversity Health System - Highland Park Hospital, Highland Park, Illinois
  - Mattoon Charleston Primary Care, Mattoon, Illinois
  - NorthShore Medical Centre, Skokie, Illinois
  - Carle Cancer Centre, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Indiana University, Indianapolis, Indiana
  - Greater Baltimore Medical Centre, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - IHA Hematology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Hospital - Brighton, Brighton, Michigan
  - IHA Hematology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Hospital- Canton, Canton, Michigan
  - IHA Hematology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Hospital - Chelsea, Chelsea, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Clinic North - Bemidji, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - St John's Hospital, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, 800 East 28th Street, Minneapolis, Minnesota
  - Hennepin County Medical Center - Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Dartmouth Hitchcock Medical Center/Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Weill Medical College of Cornell University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Einstein Campus, 1695 Eastchester Road, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, 111 East 210th Street, The Bronx, New York
  - Dickstein Cancer Treatment Centre, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Centre, Clinton, North Carolina
  - Southeastern Medical Oncology Centre, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Centre, Jacksonville, North Carolina
  - Southeastern Medical Oncology Centre, Wilson, North Carolina
  - Sanford Bismark Medical Centre, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Centre, Fargo, North Dakota
  - Sanford Medical Centre, Fargo, North Dakota
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Chagrin Highlands, Orange, Ohio
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Centre Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Centre - Sioux Falls, Sioux Falls, South Dakota
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute / University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Centre, Burlington, Vermont
  - Bon Secours Memorial Regional Medical Centre, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Centre, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- St John of God Subiaco Hospital, Perth, Western Australia, Australia
- Austria (4):
  - Univ. Klinik f. Frauenheilkunde u. Geburtshilfe, Graz
  - Univ. Klinik f. Frauenheilkunde Innsbruck, Innsbruck
  - LKH Salzburg, Salzburg
  - Med. Univ. Klinik f. Chir, Vienna
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Cliniques Universitaires Saint-Luc Brussels, Brussels
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
  - C.H.U. Sart-Tilman, Liège
  - Clinique St.Elizabeth, Namur
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver Cancer Centre, Vancouver, British Columbia
  - St Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - French Lyon Cancer Center, Lyon
  - APHP, Tenon Hospital in Paris, Paris
- Greece (2):
  - University General Hospital of Heraklion, Stavrakia, Crete
  - Laso General Hospital, First Department of Medical Oncology, Athens
- Debrecen University Dep. of Oncology, Debrecen, Hungary
- Ireland (5):
  - St Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Galway University Hospital, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (16):
  - Ospedale di Prato, Prato, Firenze
  - U.O Medicina Oncologica Ospedale di Carpi, Carpi, Modena
  - Ospedale di Trento, Trento, Trento
  - Multimedica Spa, Castellanza, Vareze
  - Centro di Riferimento Oncologico, Aviano
  - Ospedale degli Infermi - S. C. Oncologia Medica, Biella
  - Azienda Sanitaria di Bolzano, Bolzano
  - Istituto Nazionale Ricerca Cancro, Genova
  - Istituto scientifico Romagnolo per lo studio e la cura, Meldola
  - Istituto Europeo di Oncologia (IEO), Milan
  - University of Eastern Piedmont, Novara
  - Salvatore Maugeri Foundation - Medical Oncology Unit, Pavia
  - UO Oncologia, Rimini Hospital, Rimini
  - Regina Elena National Cancer Institute, Rome
  - AO Universitaria Ospedale Di Circolo e Fondazione, Varese
  - Ospedale Belcolle di Viterbo, Viterbo
- Japan (18):
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - NHO Kyushu Cancer Centre, 3-1-1 Notame Minami-ku Fukuoka-shi, Fukuoka
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - St Marianna University School of Medicine Hospital, Kawasaki
  - Kyoto University Hospital, Kyoto
  - NHO Shikoku Cancer Center, Matsuyama
  - Toranomon Hospital, Minato-ku, Tokyo
  - Kamiiida Daiichi General Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - NHO Osaka National Hospital, Ōsaka
  - Tohoku University Hospital, Sendai
  - National Cancer Center for Global Medicine, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - St Luke's International Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - University of Tsukuba, Tsukuba
- American University of Beirut Medical Center, Beirut, Lebanon
- Leiden University Medical Centre, Albinusdreef 2, Postbus 9600, Leiden, Netherlands
- Norwegian Radium Hospital (Oslo University), Oslo, Norway
- Champalimaud Cancer Center - Breast Cancer Unit, Lisbon, Portugal
- Institute of Oncology & Radiology of Serbia, Belgrade, Serbia
- Institute of Oncology Ljubljana - Medical Oncology Department, Ljubljana, Slovenia
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (18):
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Instituto Catalán de Oncología de Gerona Hospital, Girona
  - Hospital Universitario HM Sanchinarro - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Universitario Virgen del Rocio, Seville
  - Hospital Quiron Sagrado Corazon, Seville
  - Hospital Virgen De La Salud, Toledo
  - Hospital General Universitario de Valencia - Servico Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Switzerland (13):
  - Inselspital Bern, Bern, Canton of Bern
  - Spital STS AG Onkologiezentrum Thun-Berner Oberland, Thun, Canton of Bern
  - Kantonspital Baden AG, Baden
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Oncocare Bern, Bern
  - Brustzentrum Thurgau - Obstetrics and Gynecology, Frauenfeld
  - University Hospital Geneva, Geneva
  - University Hospital of Lausanne (CHUV) BH06 - Oncology Department, Lausanne
  - Brustzentum Kantonsspital St. Gallen, Sankt Gallen
  - CHCVs Hôpital de Sion - Service d'oncologie ambulatoire, Sion
  - Brust-Zentrum AG, Zurich
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] Brinton LA, Sherman ME, Carreon JD, Anderson WF. Recent trends in breast cancer among younger women in the United States. J Natl Cancer Inst. 2008 Nov 19;100(22):1643-8. doi: 10.1093/jnci/djn344. Epub 2008 Nov 11. PMID 19001605
- [Background] Leclere B, Molinie F, Tretarre B, Stracci F, Daubisse-Marliac L, Colonna M; GRELL Working Group. Trends in incidence of breast cancer among women under 40 in seven European countries: a GRELL cooperative study. Cancer Epidemiol. 2013 Oct;37(5):544-9. doi: 10.1016/j.canep.2013.05.001. Epub 2013 Jun 12. PMID 23768969
- [Background] Bentzon N, During M, Rasmussen BB, Mouridsen H, Kroman N. Prognostic effect of estrogen receptor status across age in primary breast cancer. Int J Cancer. 2008 Mar 1;122(5):1089-94. doi: 10.1002/ijc.22892. PMID 17960621
- [Background] Anders CK, Hsu DS, Broadwater G, Acharya CR, Foekens JA, Zhang Y, Wang Y, Marcom PK, Marks JR, Febbo PG, Nevins JR, Potti A, Blackwell KL. Young age at diagnosis correlates with worse prognosis and defines a subset of breast cancers with shared patterns of gene expression. J Clin Oncol. 2008 Jul 10;26(20):3324-30. doi: 10.1200/JCO.2007.14.2471. PMID 18612148
- [Derived] Demeestere I, Niman SM, Partridge AH, Diego DS, Kammler R, Ruggeri M, Colleoni M, Shimizu C, Saura C, Gelmon KA, Saetersdal AB, Kroep JR, Mailliez A, Amant F, Ruiz-Borrego M, Lee JE, Kataoka A, Walshe JM, Takei J, Borstnar S, Borges VF, Saunders C, Susnjar S, Bjelic-Radisic V, Cardoso F, Meisel JL, Kawwass JF, Spanic T, El-Abed S, Piccart M, Korde LA, Goldhirsch A, Gelber RD, Pagani O, Azim HA Jr, Peccatori FA; International Breast Cancer Study Group and the POSITIVE Trial Collaborators. Hormonal factors predictive of fertility in patients with breast cancer interrupting adjuvant endocrine therapy to attempt pregnancy in POSITIVE trial. Breast. 2025 Oct;83:104547. doi: 10.1016/j.breast.2025.104547. Epub 2025 Jul 26. PMID 40743662
- [Derived] Peccatori FA, Niman SM, Partridge AH, Ruggeri M, Colleoni M, Saura C, Shimizu C, Satersdal AB, Kroep JR, Gelmon K, Amant F, Mailliez A, Moore HCF, Ruiz-Borrego M, Walshe JM, Borges VF, Gombos A, Kataoka A, Rousset-Jablonski C, Borstnar S, Takei J, Lee JE, Saunders C, Bjelic-Radisic V, Susnjar S, Cardoso F, Klar NJ, Ferreiro T, El-Abed S, Piccart M, Korde LA, Goldhirsch A, Gelber RD, Pagani O, Azim HA Jr; International Breast Cancer Study Group and the POSITIVE Trial Collaborators. Breastfeeding After Hormone Receptor-Positive Breast Cancer: Results From the POSITIVE Trial. J Clin Oncol. 2025 Aug 20;43(24):2712-2719. doi: 10.1200/JCO-24-02697. Epub 2025 Jul 9. PMID 40632989
- [Derived] Partridge AH, Niman SM, Ruggeri M, Peccatori FA, Azim HA Jr, Colleoni M, Saura C, Shimizu C, Saetersdal AB, Kroep JR, Mailliez A, Warner E, Borges VF, Amant F, Gombos A, Kataoka A, Rousset-Jablonski C, Borstnar S, Takei J, Lee JE, Walshe JM, Ruiz-Borrego M, Moore HCF, Saunders C, Bjelic-Radisic V, Susnjar S, Cardoso F, Smith KL, Ferreiro T, Ribi K, Ruddy K, Kammler R, El-Abed S, Viale G, Piccart M, Korde LA, Goldhirsch A, Gelber RD, Pagani O; International Breast Cancer Study Group; POSITIVE Trial Collaborators. Interrupting Endocrine Therapy to Attempt Pregnancy after Breast Cancer. N Engl J Med. 2023 May 4;388(18):1645-1656. doi: 10.1056/NEJMoa2212856. PMID 37133584
- [Derived] Perachino M, Poggio F, Arecco L, Blondeaux E, Spinaci S, Marrocco C, Levaggi A, Lambertini M. Update on Pregnancy Following Breast Cancer Diagnosis and Treatment. Cancer J. 2022 May-Jun 01;28(3):176-182. doi: 10.1097/PPO.0000000000000599. PMID 35594464